CLINICAL TRIAL: NCT04985214
Title: Assessment of the Quality of Life of Patients With Lymphomas Treated With Oral Therapy
Acronym: EVEREST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0465
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Quality of Life
Keywords: oral therapy; lymphoma; quality of life
MeSH Terms: conditions — Lymphoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oral therapy: Patients included in the PK-E3i clinical study or patients with hemopathies starting treatment with oral therapy.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire on the quality of life

SUMMARY:
The emergence of new anti-cancer drugs orally administered has revolutionized the prognosis and modalities of management of several lymphomas over the past decade. Today, half of patients receive oral therapy at home. Ibrutinib, acalabrutinib, idelalisib, venetoclax and lenalidomide are oral therapies used in the treatment of Chronic Lymphoid Leukemia, Follicular Lymphoma, Waldenström's disease and mantle cell lymphoma, in relapsing but soon to be 1st line.

Nevertheless, clinical trials leading to marketing authorizations for these drugs were performed in a small number of patients and very little data is available on their use in real life conditions. Their impact on the quality of life of patients also remains to be assessed.

The aim of this clinical research is to evaluate quality of life of patients at the initiation of the first oral therapy and every year for 5 years. This study will also identify factors (biological and non-biological: quality of life, shared decision-making ...) associated with a good response of patients and follow-up for the occurrence of long-term adverse reactions (5 years).

DETAILED DESCRIPTION:
Prospective longitudinal cohort. This observational study is monocentric. For each patient, data will be collected during 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the PK-E3i clinical study OR
* Over the age of 18
* Patients with hemopathies and starting treatment with oral therapy (idelalisib, ibrutinib, venetoclax, lenalidomide, acalabrutinib…)
* Be able to understand the objective and the constraints related to research
* Patient having read the information notice and the non-objection form
* Social Security affiliation

Exclusion Criteria:

* Pregnant women
* Persons under legal protection of adults
* Patients under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hemopathies and starting treatment with oral therapy (idelalisib, ibrutinib, venetoclax, lenalidomide, acalabrutinib…)
Sampling Method: Non-Probability Sample
Enrollment: 464 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life measurement | 5 years
  Evaluation of the quality of life score, throught the quality of life scale (higher score associated with poor quality of life)

SECONDARY OUTCOMES:
Evaluation of patients factors | 5 years
  Collect of clinical and socio-professional characteristics of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Loïc YSEBAERT, Prof., Principal Investigator — University Hospital, Toulouse
Locations (14):
- France (14):
  - CH de Bayonne, Bayonne
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - CH Versailles, Le Chesnay
  - CH Le Mans, Le Mans
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nîmes, Nîmes
  - CH de Perpignan, Perpignan
  - Hospices Civils de Lyon, Pierre-Bénite
  - Loïc YSEBAERT, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No